CLINICAL TRIAL: NCT04714541
Title: Case Series: A Sequenced Treatment Using a Modified Ketogenic Diet and Ketamine for Severe and Enduring Anorexia Nervosa
Brief Title: Modified Ketogenic Diet and Ketamine for Anorexia Nervosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Homeostasis Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-2020 ANKK
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: The 5 Participants Undergo A Sequenced Treatment of Adopting A Ketogenic Diet For at Least 4 Weeks, Followed by A Series of Intravenous Ketamine Infusions
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet Adoption Followed by Ketamine Infusion (Experimental): All 5 Participants Will Be Educated to Adopt a Ketogenic Diet, As Outpatient. After at Least 4 Weeks on the Diet, They Will Have A Series of Titrated Intravenous Ketamine Infusions Over A 2 Week Period
  Interventions: Drug: Ketamine Hcl 50Mg/Ml Inj

INTERVENTIONS:
Drug: Ketamine Hcl 50Mg/Ml Inj — Racemic Ketamine Will Be Infused At A Starting Dose of 0.75 mg/kg Over A Period of 45 Minutes. The Dose Will be Titrated, Based on Clinical Signs With Changes of 0.3mg/kg Up to Maximum of 0.95 mg/kg, and Lowest Dose of 0.3 mg/kg

SUMMARY:
This Open-Label Pilot Study Aims to Determine Whether a Two-Part Sequenced Out Patient Procedure Utilizing a Modified Ketogenic Diet Followed by a Series of Titrated Ketamine Infusions Results in Improvement or Remission of Chronic Anorexia Nervosa in Adults with Symptoms of Anorexia for at Least 3 Years Despite Treatment Involving at Least 2 Different Modalities. The Hypothesis is That the Diet Addresses Core Metabolic Deficits in the "Anorexic Brain" and Primes the Response to Ketamine.

DETAILED DESCRIPTION:
Participants Who Are Deemed Eligible Will Participate in an Open-Label Clinical Trial Using a Sequenced Treatment Previously Reported in One Case Study to Result in Complete and Sustained Remission of Anorexia Nervosa for Over One Year (and Continuing).

Part 1 Involves a Group 2-Day Immersive In-Person Educational Program to Begin a Modified Ketogenic Diet, Under the Supervision of a Nutritionist Who Has Decades of Experience in Designing Ketogenic Diets for Seizure Patients. This Group Experience is Followed by a 4 Week Period of At-Home Adoption of the Diet, With Close Phone and E-Mail Follow-up.

Part 2 Involves Administration of a Series of Titrated Intravenous Ketamine Infusions Scheduled Over 2 Weeks.

During Part 1, and Part 2, There Will Be a Range of Objective and Psychological Measures To Assess Safety and Response. The Participants Will be Followed For 12 Months.

ELIGIBILITY:
Inclusion Criteria:

* Adults Between 18 and 65
* Anorexia Nervosa Diagnosis For at Least 3 Years
* Treatment Resistance, as Evidenced by Having Failed at Least 2 Treatments
* Body Mass Index (BMI) Greater than or Equal to 18.5
* Stable Weight for the Last 3 Months (No Consistent Change Greater than 5 Pounds)
* Abstinence From Substance Abuse for At Least 3 Months
* No Cannabis Use for At Least 3 Months
* Currently Under the Care of a Primary Care Provider (PCP)
* Participant Must Agree to have PCP Contacted by Study Staff
* Willingness to Participant in a 2-Day Program in Central Connecticut
* Identified Support Partner Who Will Attend Program
* Willingness to Have Weight Recorded and Reported by PCP or Support Partner
* Willingness to Attend 4-6 Clinic Visits For Ketamine Infusion
* Willingness to Be Contacted for Follow Up for 12 Months
* Willingness to Abide By All COVID Safety Measures

Exclusion Criteria

* Concomitant Disease (Gastroentestinal, Renal, Respiratory, Cardiac, Etc) or Any Clinically Significant Finding at Screening that Would Pose a Risk to the Participant
* Primary Carnitine Deficiency, Beta Oxidation Defects, Pyruvate Carboxylase Deficiency, Porphyria, or Treatment with Carbonic Anhydrase Inhibitors
* Bulimia Nervosa as The Primary Diagnosis
* Weight Change of Greater Than 5 Pounds in Last 3 Months
* Pregnancy
* Sexually Active Females Not Using Birth Control
* Interstitial Cystitis
* Unmanaged/Unstable Hypertenison (Greater than 140 Systolic; 90 Diastolic
* Cardiac Arrythmia
* Uncontrolled Seizure Disorder or Seizure Withen 30 Days Prior to Screening
* QTc Interval of 470 ms or Greater
* Current or Past History of Psychotic Disorder
* Active Suicidal Ideation
* Enrolled in any Clinical Trial or Used Any Investigational Agent, Device, and/or Investigational Procedure Within 30 Days Before Screening, or Does so Concurrently With this Study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Changes in Eating Disorder Examination Questionnaire (EDE-Q) Score | Change from Baseline at 4 weeks; 8 Weeks; 3 Months; 6 Months; 9 Months; 12 Months
  A 28-item Self Report Scale that Assesses the Range and Severity of ED symptoms
Change in Eating Disorder Recovery Endorsement Questionnaire (EDREQ) Score | Change from Baseline at 4 Weeks, 8 Weeks, 3 Months; 6 Months, 9 Months, 12 Months
  Self Report Scale that Assesses The Indicators of Recovery
Change in Clinical Impairment Assessment (CIA) For Eating Disorders Scale | Change from Baseline at 4 Weeks; 8 Weeks; 3 Months; 6 Months; 9 Months;12 Months
  A 16-Item Self Administered Rating Scale Which Measures PsychoSocial Impairment
Change in Behavior and Mood and Thinking as Measured by Interview | Change from Baseline at 4 Weeks, 8 Weeks, 3 Months, 6 Months, 9 Months, 12 Months
  Qualitative Analysis of Research- Associate Administered Questionnaire

SECONDARY OUTCOMES:
Change in Body Weight/Body Mass Index | Change from Baseline Biweekly for Weeks 1,2,3, and 4, Weekly for weeks 5,6,7,8.then 3 Months, 6 Months, 9 Months, 12 Months s and Prior to Every Ketamine Infusion 8 Weeks; 3 Months; 6 Months; 9 Months;12 Months
  Weight to Be Measured By Local Clinician or Support Person to Ensure Safety

OTHER OUTCOMES:
Breath Acetone Measure | Change from Baseline Daily Week 1,2,3, and 4 ,8 Weeks, 3 Months, 6 Months, 9 Months, 12 Months
  Acetone Measured by Participant with Portable Breath Acetone Meter
Brief 24- Hour Food Recall | Change from Baseline Weeks1,2,3,4 then, 8 Weeks, 3 Months, 6 Months, 9 Months 12 Months
  Obtained by Research Associate
Change in Food Preference as Assessed by The Geiselman Food Preference Questionnaire | Change from Baseline at 4 Weeks, 8 Weeks, then 3 Months, 6 Months, 9 Months 12 Months
  Self Administered Questionnaire
Change in Depressive Symptoms as Assessed by Patient Health Questionnaire | Change from Baseline at Week 4, 5, 6, and 3 Months, 6 Months, 9 Months 12 Mos
  A 9 Item Self Administered Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lori Calabrese, MD, Principal Investigator — Innovative Psychiatry So Windsor; Lori Calabrese, MD, Principal Investigator — Innovative Psychiatry, So Windsor
Locations (1):
- Lori Calabrese MD Innovative Psychiatry, South Windsor, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No